CLINICAL TRIAL: NCT00036296
Title: Effects of Talampanel on Patients With Advanced Parkinson's Disease Who Have Been on Sinemet for More Than 5 Years and Have Dyskinesia (Abnormal Involuntary Movements)
Brief Title: Effects of Talampanel on Patients With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Rivka Kreitman, Ph.D., Vice President, Innovative Research and Development, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXL-202-18-189
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2009-10

CONDITIONS: Dyskinesias; Parkinson Disease; Movement Disorders
Keywords: Involuntary Movements; Abnormal Movements; Advanced Parkinson's disease; Levodopa induced dyskinesia
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Movement Disorders | interventions — talampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 75mg per day (in 3 doses) Talampanel for 22 days
  Interventions: Drug: talampanel
- 2 (Placebo Comparator): 3 doses a day for 22 days
  Interventions: Drug: talampanel

INTERVENTIONS:
Drug: talampanel — 75mg per day divided into 3 doses for 22 days

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the study drug, Talampanel, when used to treat patients with involuntary movements known as dyskinesias, as a result of treatment to Parkinson's disease.

It is not clear why people with Parkinson's disease develop involuntary movements (dyskinesias) but studies show that blocking receptors in the brain for a chemical called glutamate decreases these movements. Talampanel is a drug which blocks these receptors.

ELIGIBILITY:
Inclusion Criteria:

* Troublesome on-period dyskinesias as defined by a Unified Parkinson's Disease Rating Scale (UPDRS) dyskinesia sub-score >25% of Duration of dyskinesia during waking hours and 33 must have moderate disability
* Lang-Fahn dyskinesia rating score more than 2 for at least two of the 5 tasks
* Must have Dyskinesia on average 25% of waking hours/day based on Patient Diaries
* Have been diagnosed with Parkinson's disease > 5 years at Screening

Exclusion Criteria:

* Previous surgical therapies for PD
* Isolated or predominantly diphasic dyskinesias
* Moderate Dementia
* On disallowed concomitant medications including CYP3A4 inhibitors and inducers, amantadine, etc.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)